CLINICAL TRIAL: NCT07206966
Title: Validation of the Swedish Translation of a Brief Shame Measure, the External and Internal Shame Scale (EISS)
Brief Title: Validation of the Swedish Translation of a Brief Shame Measure, the External and Internal Shame Scale
Acronym: EMBER-1
Status: Not yet recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: EMBER-1
Record Dates: First submitted 2025-09-15; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Shame
Keywords: Psychometrics; Psychological Tests; Shame; Patient Health Questionnaire; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- General Population: Participants Recruited through Social Media
- Women Subjected to Intimate Partner Violence/Sexual Assault: Patients at the NCK Outpatient Clinic at Uppsala University Hospital
- Cardiology Patients: Patients at the Cardiology Outpatient Clinic at Uppsala University Hospital
- Patients with Excessive Daytime Sleepiness: Patients at the Outpatient Sleep Clinic at Uppsala University Hospital

SUMMARY:
Shame is a normal emotion that people sometimes have. Experiencing a lot of shame has however been found to have a link to ill mental and somatic health. Therefore it is of interest to have a brief way of measuring shame. External and Internal shame scale (EISS) is a questionnaire with 8 items that is available in several languages, but not yet in Swedish. The researchers have translated it to Swedish and will investigate how well the Swedish version works for measuring shame. 300 participants are enrolled via social media and asked to complete the EISS as well as two other scales for comparison. Participants are also asked about their age and gender. In addition, a total of 150 participants will be recruited from 3 outpatient clinics in order to check how the scale works in clinical settings. The researchers will use the answers to statistically calculate the scientific properties of the EISS.

ELIGIBILITY:
Inclusion Criteria

* Must be 18 years of age or above
* Must be capable of communicating in Swedish
* Participants in clinical samples must be patients at one of the clinics involved in the study.

Exclusion criteria

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample + clinical samples from 3 outpatient clinics at Uppsala University Hospital: the NCK Outpatient Clinic, the Cardiology Outpatient Clinic and the Outpatient Sleep clinic.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
EISS | Within a week of enrollment
  External and Internal Shame Scale, an 8-item measure with a total scale ranging from 0 to 32 points, and two subscales of internal and external shame, ranging from 0 to 16 each. Self-assessment of how often one feels what is described in each item, ranging from "never" (0) to "always" (4).

SECONDARY OUTCOMES:
ISS | Within a week of enrollment
  Internalized Shame Scale consists of 30 items, of which 24 measure internalized shame and 6 measure self esteem. Self assessment of "how often one feels or experiences" each of the items, ranging from "never" (0) to "almost always" (4).
PHQ-9 | Within a week of enrollment
  Patient Health Questionnaire - 9 item version is a widely used depression screening tool, measuring levels of depression symptoms. Self-assessment of how often one has been bothered by the symptoms in question over the past 2 weeks, ranging from "not at all" (0) to "nearly every day" (3). Total range 0-27.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Överlien, professor, Principal Investigator — The National Centre for Knowledge on Men's Violence Against Women, Uppsala university
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No